CLINICAL TRIAL: NCT04011722
Title: Evaluation of the Portico™ NG (Next Generation) Transcatheter Aortic Valve in High and Extreme Risk Patients With Symptomatic Severe Aortic Stenosis
Brief Title: Portico Next Generation Approval Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10297; ABT-CIP-10308 (Other: Abbott)
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Symptomatic Severe Aortic Stenosis
Keywords: Aortic Stenosis; Transcatheter Aortic Valve Implantation; Heart Valve Disease; High Surgical Risk; Portico NG (Navitor) Valve; Extreme Surgical Risk; Navitor Titan Valve
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Devices under investigation in this clinical study include the Portico™ (Navitor) Valve (23mm, 25mm, 27mm and 29mm sizes), Navitor Titan Valve (35 mm), FlexNav™ Delivery System (small and large) and Portico™ NG (Navitor) Loading System(s) (small and large), and Navitor Loading System - LG+, all of which are currently approved for investigational use only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Portico™ NG (Navitor) valve, FlexNav™ Delivery System (Experimental): Portico ™ NG (Navitor) valve implantation with the new generation Portico NG (Navitor) valve (23mm, 25mm, 27mm and 29mm sizes), and the second-generation FlexNav Delivery system (small and large), Portico™ NG (Navitor) Loading System(s) (small and large).
  Interventions: Device: Portico™ NG (Navitor) Valve and FlexNav™ Delivery System
- Navitor Titan Valve (Experimental): Navitor Titan Valve (35mm) implantation with the large FlexNav Delivery system and Navitor Loading System - LG+.
  Interventions: Device: Navitor Titan Valve (35mm) Valve and Large FlexNav™ Delivery System

INTERVENTIONS:
Device: Portico™ NG (Navitor) Valve and FlexNav™ Delivery System — Subjects will undergo transcatheter aortic valve implantation (TAVI) with the new generation Portico NG (Navitor) valve and second-generation FlexNav Delivery system via a transfemoral or alternative access approach according to the site's anesthesia protocol for TAVR procedures.
  Arms: Portico™ NG (Navitor) valve, FlexNav™ Delivery System
Device: Navitor Titan Valve (35mm) Valve and Large FlexNav™ Delivery System — Subjects will undergo transcatheter aortic valve implantation (TAVI) with the Navitor Titan valve and large FlexNav Delivery system via a transfemoral or alternative access approach according to the site's anesthesia protocol for TAVR procedures.
  Arms: Navitor Titan Valve

SUMMARY:
The purpose of this clinical study is to evaluate the acute safety and effectiveness of the next-generation Navitor (Portico™ NG) Transcatheter Aortic Heart Valve as assessed by the rate of all-cause mortality at 30 days and the rate of moderate or greater paravalvular leak at 30 days in a high or extreme surgical risk patient population to support CE (Conformité Européenne) Mark and FDA approval.

DETAILED DESCRIPTION:
The Portico NG Approval study will be conducted as a prospective, multi-center, international, single-arm investigational study.

Up to 399 (includes up to 20 roll-ins) high or extreme risk patients with symptomatic, severe native aortic stenosis who are determined by an independent subject selection committee to meet eligibility criteria for Navitor Transcatheter Aortic Heart Valve implantation will undergo Navitor Valve implantation via a transfemoral or alternative access approach according to the site's anesthesia protocol for TAVR (transcatheter aortic valve replacement) procedure.

Subjects participating in the clinical study will be followed for a total of 12 months with data collected at screening, baseline, procedure, prior to hospital discharge, and follow-up at 30 days, 12 months and annually at 2, 3, 4 and 5 years.

This study will also include a product size extension, Navitor Titan™ valve, which includes up to 90 subjects (Titan cohort) who will undergo an implant attempt with the Navitor Titan valve. Subjects enrolled in the Titan cohort will undergo the same screening, baseline, procedure and follow-up assessments as the Portico NG cohort.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects must have a Society of Thoracic Surgeons (STS) score of ≥7% OR documented heart team agreement of high or extreme risk for surgical aortic valve replacement due to frailty or co-morbidities not captured by the STS score.
2. Subject has symptomatic aortic stenosis as demonstrated by NYHA (New York Heart Association) Functional Classification of II, III, or IV.
3. Subject has senile degenerative aortic valve stenosis with echo-derived criteria, defined as: aortic valve area (AVA) of ≤ 1.0 cm2 (or indexed EOA (effective orifice area) ≤ 0.6 cm2/m2) AND mean gradient ≥40 mmHg or peak jet velocity ≥ 4.0 m/s or doppler velocity index (DVI) ≤0.25. (Qualifying AVA baseline measurement must be within 90 days prior to informed consent).
4. Aortic annulus diameter of 19-30mm and ascending aorta diameter for the specified valve size listed in the IFU (Instructions For Use), as measured by CT (Computed Tomography)

Key Exclusion Criteria:

1. Evidence of an acute myocardial infarction (defined as: ST Segment Elevation as evidenced on 12 Lead ECG) within 30 days prior to index procedure.
2. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to index procedure.
3. Blood dyscrasias as defined: leukopenia (WBC<3000 mm3), acute anemia (Hb < 9 g/dL), thrombocytopenia (platelet count <50,000 cells/mm³). History of bleeding diathesis or coagulopathy
4. Active peptic ulcer or upper GI bleeding within 3 months prior to index procedure that would preclude anticoagulation
5. Recent (within 6 months prior to index procedure date) cerebrovascular accident (CVA) or a transient ischemic attack (TIA).
6. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation 3-4+).
7. Pre-existing prosthetic heart valve or other implant in any valve position, prosthetic ring, severe circumferential mitral annular calcification (MAC) which is continuous with calcium in the left ventricular outflow tract (LVOT), severe (greater than or equal to 3+) mitral insufficiency, or severe mitral stenosis with pulmonary compromise.
8. Minimum access vessel diameter of <5.0mm for small FlexNav™ Delivery System and <5.5 mm for large FlexNav™ Delivery System

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (21):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Atlantic Health System - Morristown Memorial Hospital, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Montefiore Medical Center - Moses Division, New York, New York
  - Mission Health & Hospitals, Asheville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - The Methodist Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain St. George Regional Hospital, St. George, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Australia (3):
  - St. Andrew's Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Rigshospitalet, Copenhagen, Denmark
- Policlinico San Donato, San Donato Milanese, Lombard, Italy
- United Kingdom (2):
  - Royal Victoria Hospital, Belfast, Northern Ireland
  - Morriston Hospital - ABM University Health Board, Morriston, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reardon MJ, Chehab B, Smith D, Walton AS, Worthley SG, Manoharan G, Sultan I, Yong G, Harrington K, Mahoney P, Kleiman N, Makkar RR, Fontana G, DeLago A, Ramana RK, Bates N, Sondergaard L. 30-Day Clinical Outcomes of a Self-Expanding Transcatheter Aortic Valve: The International PORTICO NG Study. JACC Cardiovasc Interv. 2023 Mar 27;16(6):681-689. doi: 10.1016/j.jcin.2023.02.002. Epub 2023 Feb 27. PMID 36990558

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
Started | 260 | 73
Completed | 260 | 73
Not Completed | 0 | 0
Period: Procedure
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
Started | 260 | 73
Completed | 260 | 73
Not Completed | 0 | 0
Period: Discharge
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
Started | 260 | 73
Completed | 260 | 73
Not Completed | 0 | 0
Period: 30 Days
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
Started | 260 | 73
Completed | 255 | 72
Not Completed | 5 | 1
Not completed — Death | 5 | 1
Period: 1 Year
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
Started | 255 | 72
Completed | 228 | 44
Not Completed | 27 | 28
Not completed — Death | 13 | 5
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Missed Visit | 6 | 1
Not completed — Pending Visit | 0 | 11
Not completed — Not Yet Due | 0 | 9
Period: 2 Year
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
Started | 234 (At 2 years, number of subjects started is 234 (228(1 yr completed) + 6 (missed 1 year visit)).) | 64 (Not all subjects completed the 1 yr visit. Hence the number of participants to start a Period is not equal to the number who completed previous Period.)
Completed | 155 | 5
Not Completed | 79 | 59
Not completed — Death | 16 | 1
Not completed — Withdrawal by Subject | 10 | 1
Not completed — Missed Visit | 9 | 0
Not completed — Visit Pending | 1 | 3
Not completed — Not Yet Due | 43 | 54
Period: 3 Year
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
Started | 208 (Not all subjects completed the 2 yr visit. Hence the number of participants to start a Period is not equal to the number who completed previous Period.) | 0 (Navitor Titan Cohort is yet to complete 3 years follow-up visits)
Completed | 61 | 0
Not Completed | 147 | 0
Not completed — Death | 10 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Missed Visit | 2 | 0
Not completed — Pending Visit | 34 | 0
Not completed — Not Yet Due | 99 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve | Total
Number analyzed (Participants) | 260 | 73 | 333
Age, Continuous [Mean (Standard Deviation); unit: Years] | 83.4 (5.4) | 80.6 (5.2) | 82.0 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 1 | 150
  Male | 111 | 72 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 257 | 71 | 328
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 189 | 56 | 245
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 64 | 16 | 80
NYHA Class [Count of Participants; unit: Participants] — (NYHA CLASS) Class I: cardiac disease but without resulting limitations of physical activity.
  Class II: cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest.
  Class III: cardiac disease resulting in marked limitation of physical activity. Patients are comfortable at rest.
  Class IV: cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
  Participants
    NYHA I | 0 | 0 | 0
    NYHA II | 117 | 53 | 170
    NYHA III | 138 | 19 | 157
    NYHA IV | 5 | 1 | 6
STS Risk of Mortality [Mean (Standard Deviation); unit: Percentage of Risk] — The Society of Thoracic Surgeons (STS) Risk Score is a model that predicts the risk of surgical mortality for open heart surgery. The score is based on data from the STS National Adult Cardiac Surgery Database and uses a multivariable logistic regression model to calculate predicted probabilities ranging from 0 to 1. The STS score classifies patients into three risk groups based on their predicted risk of mortality:
  Low risk: Less than 4% Intermediate risk: 4-8% High risk: 8% or greater
  Percentage of Risk | 3.9 (2.1) | 2.7 (1.3) | 3.3 (1.7)
EuroSCORE II [Mean (Standard Deviation); unit: Percentage of Risk] — EuroSCORE II estimates the 30-day mortality risk after cardiac surgery, expressed as a percentage. EuroSCORE II score has three groups, 1. low risk defined as EuroSCORE < 4%, 2. intermediate risk as 4-8%, and 3. high risk as > 8%.
  Percentage of Risk | 3.4 (2.3) | 2.7 (1.7) | 3.05 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint is All-cause Mortality
Description: All-cause mortality is defined as the total number of deaths in each cohort at 30 days.
Time Frame: at 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
Number analyzed (Participants) | 260 | 73
Participants | 5 | 1

2. Primary Outcome: Primary Effectiveness Endpoint is Moderate or Greater Paravalvular Leak
Description: Number of participants with moderate or greater paravalvular leak at 30 days.
Time Frame: at 30 days
Population: All available subjects with echocardiographic data have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
Number analyzed (Participants) | 248 | 68
Participants
  None/Trace PVL | 198 | 61
  Mild PVL | 50 | 7
  Moderate PVL | 0 | 0
  Severe PVL | 0 | 0

3. Secondary Outcome: Non-hierarchical Composite of All-cause Mortality, Disabling Stroke, Life Threatening Bleeding, Acute Kidney Injury (Stage 3), or Major Vascular Complications
Description: The secondary endpoint is defined as a non-hierarchical composite of all-cause mortality, disabling stroke, life threatening bleeding, acute kidney injury (stage 3), or major vascular complications at 30 days.
Time Frame: at 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
Number analyzed (Participants) | 260 | 73
Participants
  All-Cause Mortality | 5 | 1
  Myocardial Infarction | 2 | 1
  All Stroke | 10 | 2
  Transient Ischemic Attack | 2 | 2
  Life-Threatening Bleeding | 10 | 0
  Major Bleeding | 12 | 2
  Major Vascular Complications | 11 | 3
  Acute Kidney Injury | 5 | 0
  Valve Thrombosis | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events through 3 year follow-up visit.
Arm/Group | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System | Navitor Titan Valve
All-Cause Mortality (participants affected / at risk) | 44/260 | 6/73
Serious Adverse Events (participants affected / at risk) | 180/260 | 50/73
Other Adverse Events (participants affected / at risk) | 197/260 | 54/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System (N=260) | Navitor Titan Valve (N=73)
Angina Pectoris (Cardiac disorders) | 13 (17) | 2 (2)
Aortic Dissection (Cardiac disorders) | 1 (1) | 1 (1)
Aortic Aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmias (Cardiac disorders) | 26 (34) | 7 (8)
Arterial Hypertension (Cardiac disorders) | 6 (6) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 4 (4) | 2 (2)
Cardiac Perforation (Cardiac disorders) | 2 (2) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0)
EKG Finding (Cardiac disorders) | 6 (6) | 2 (2)
Echo Finding (Cardiac disorders) | 3 (3) | 1 (2)
Endocarditis (Cardiac disorders) | 4 (4) | 0 (0)
General - Cardiovascular Symptoms (Cardiac disorders) | 1 (1) | 0 (0)
Heart Block (Cardiac disorders) | 49 (49) | 24 (25)
AV Block (Cardiac disorders) | 3 (3) | 0 (0)
First Degree Heart/AV Block/Cardiac Arrhythmia - 1st degree AV Block (Cardiac disorders) | 3 (3) | 3 (3)
Heart Block (Cardiac disorders) | 2 (2) | 2 (2)
Left Bundle Branch Block/Complete Left Bundle Branch Block (Cardiac disorders) | 10 (10) | 7 (7)
Mobitz II Block (Cardiac disorders) | 1 (1) | 1 (1)
Right Bundle Branch Block/Complete Right Bundle Branch Block (Cardiac disorders) | 2 (2) | 1 (1)
Third Degree Heart Block (Complete Heart Block) (Cardiac disorders) | 28 (28) | 11 (11)
Heart Failure (Cardiac disorders) | 23 (31) | 9 (12)
Heart Murmur (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 14 (14) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 7 (7) | 0 (0)
Myocardial Ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 5 (5) | 0 (0)
Pericardial Tamponade (Cardiac disorders) | 3 (3) | 0 (0)
Pulmonary Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Shock (Cardiac disorders) | 1 (1) | 0 (0)
Valve (Cardiac disorders) | 7 (9) | 1 (1)
Benign Tumors (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Skin Cancer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nose and Paranasal Sinuses (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanic Membrane and Ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dehydration (Endocrine disorders) | 3 (3) | 1 (1)
Disorders of Carbohydrate Metabolism (Endocrine disorders) | 6 (6) | 1 (1)
Hyperkalemia (Endocrine disorders) | 3 (3) | 0 (0)
Hypernatremia (Endocrine disorders) | 1 (1) | 0 (0)
Hypokalemia (Endocrine disorders) | 3 (3) | 1 (1)
Hyponatremia (Endocrine disorders) | 2 (2) | 2 (2)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel Obstruction (Gastrointestinal disorders) | 3 (4) | 0 (0)
Colon Polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 10 (13) | 3 (3)
Hepatic and Biliary Disorders (Gastrointestinal disorders) | 5 (9) | 2 (2)
Hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Melena (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Tumors (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 13 (14) | 7 (8)
Hematuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Prostate Disease (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal Failure (Renal and urinary disorders) | 6 (6) | 0 (0)
Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 6 (7) | 1 (1)
Urinary Tract Infections (Renal and urinary disorders) | 11 (15) | 3 (5)
Breast Cancer (General disorders) | 1 (1) | 0 (0)
Abnormal Lab Value (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Anemias (Blood and lymphatic system disorders) | 15 (19) | 3 (3)
Bacteremia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Bleeding (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Blood Loss (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Deep Vein/Venous Thrombosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukemias (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 2 (2)
Thrombus (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Bacterial Infections (Infections and infestations) | 2 (2) | 0 (0)
C. Difficile Infection (Infections and infestations) | 1 (1) | 1 (1)
Miscellaneous Infections (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 9 (9) | 1 (1)
Septicemia (Infections and infestations) | 1 (1) | 0 (0)
Cancer (Injury, poisoning and procedural complications) | 10 (12) | 0 (0)
Claudication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device/Delivery System (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Emesis/Vomiting (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 17 (20) | 0 (0)
Fever (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Lacerations (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Non-Study Procedure Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other (Injury, poisoning and procedural complications) | 48 (61) | 0 (0)
Swelling (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Dissection (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Weakness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 8 (9) | 2 (3)
General - Musculoskeletal Symptoms (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Osteoarthritis/Degenerative Joint Disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Cord Disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Toe Inflammation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Arteriovenous Malformation (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carpal Tunnel (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Nervous system disorders) | 2 (2) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 2 (2)
General - Neurological Symptoms (Nervous system disorders) | 3 (3) | 1 (1)
Hemiparesis/Weakness (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Neurological Hematoma (Nervous system disorders) | 3 (4) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1)
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 15 (16) | 3 (3)
Syncope (Nervous system disorders) | 9 (10) | 1 (1)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 7 (11) | 2 (2)
Vaso Vagal Response (Nervous system disorders) | 1 (1) | 2 (2)
Macular Degeneration (Eye disorders) | 1 (1) | 0 (0)
Chronic Obstructive Airway Disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypersensitivity Diseases of the Lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Disorders (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 4 (4)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 4 (6)
Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheeze (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
VASC Bleeding (Vascular disorders) | 4 (5) | 1 (1)
VASC Hematoma (Vascular disorders) | 1 (1) | 0 (0)
VASC Pseudoaneurysm (Vascular disorders) | 4 (4) | 0 (0)
VASC Vessel Perforation (Vascular disorders) | 2 (2) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cancer (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Device/Delivery System (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Elective Procedure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Fever (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Other (Injury, poisoning and procedural complications) | 0 (0) | 16 (26)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Portico™ NG (Navitor) Valve, FlexNav™ Delivery System (N=260) | Navitor Titan Valve (N=73)
Angina Pectoris (Cardiac disorders) | 11 (11) | 0 (0)
Arrhythmias (Cardiac disorders) | 30 (32) | 9 (9)
Arterial Hypertension (Cardiac disorders) | 19 (20) | 1 (1)
EKG Finding (Cardiac disorders) | 8 (8) | 2 (2)
Echo Finding (Cardiac disorders) | 1 (1) | 1 (1)
General - Cardiovascular Symptoms (Cardiac disorders) | 2 (2) | 1 (1)
Heart Block (Cardiac disorders) | 60 (71) | 15 (17)
AV Block (Cardiac disorders) | 1 (1) | 0 (0)
First Degree Heart/AV Block/Cardiac Arrhythmia - 1st degree AV Block (Cardiac disorders) | 12 (12) | 2 (2)
Heart Block (Cardiac disorders) | 1 (1) | 0 (0)
High Grade Block/Advanced AV Block (Cardiac disorders) | 1 (1) | 0 (0)
Incomplete Left Bundle Branch Block (Cardiac disorders) | 1 (1) | 0 (0)
Left Bundle Branch Block/Complete Left Bundle Branch Block (Cardiac disorders) | 49 (50) | 13 (13)
Right Bundle Branch Block/Complete Right Bundle Branch Block (Cardiac disorders) | 1 (1) | 1 (1)
Second Degree Heart Block (Cardiac disorders) | 1 (1) | 1 (1)
Third Degree Heart Block (Complete Heart Block) (Cardiac disorders) | 3 (3) | 0 (0)
Heart Failure (Cardiac disorders) | 16 (16) | 4 (5)
Hypertensive Crisis (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 13 (13) | 5 (6)
Myocardial Infarction (Cardiac disorders) | 3 (4) | 1 (1)
Myocardial Ischemia (Cardiac disorders) | 3 (3) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 2 (2) | 0 (0)
Pulmonary Hypertension (Cardiac disorders) | 4 (4) | 1 (1)
Sinus Node Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Valve (Cardiac disorders) | 1 (1) | 1 (1)
Abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Contusion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Disorders of Cornification (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dental Disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Nose and Paranasal Sinuses (Ear and labyrinth disorders) | 4 (4) | 0 (0)
Tympanic Membrane and Ear (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Disorders of Carbohydrate Metabolism (Endocrine disorders) | 4 (4) | 1 (1)
Hyperkalemia (Endocrine disorders) | 1 (1) | 0 (0)
Hypernatremia (Endocrine disorders) | 1 (1) | 0 (0)
Hypokalemia (Endocrine disorders) | 4 (4) | 1 (1)
Hyponatremia (Endocrine disorders) | 4 (4) | 1 (1)
Thyroid Disorders (Endocrine disorders) | 4 (4) | 0 (0)
Colon Polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (8) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhoids/Piles (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic and Biliary Disorders (Gastrointestinal disorders) | 2 (2) | 0 (0)
Acute Kidney Injury (General disorders) | 12 (13) | 1 (1)
Dysuria (General disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 5 (6) | 1 (1)
Hematuria (General disorders) | 1 (1) | 0 (0)
Prostate Disease (General disorders) | 2 (2) | 0 (0)
Renal Insufficiency (General disorders) | 2 (2) | 0 (0)
Urinary Retention (General disorders) | 4 (4) | 2 (2)
Urinary Tract Infections (General disorders) | 15 (16) | 3 (4)
Breast Cancer (General disorders) | 1 (1) | 0 (0)
Abnormal Lab Value (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Anemias (Blood and lymphatic system disorders) | 15 (15) | 8 (8)
Bleeding (Blood and lymphatic system disorders) | 5 (6) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 12 (13) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (12) | 4 (4)
Thrombus (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bacterial Infections (Infections and infestations) | 1 (1) | 0 (0)
C. Difficile Infection (Infections and infestations) | 1 (2) | 1 (1)
Viral (Infections and infestations) | 10 (10) | 0 (0)
Cancer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Claudication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device/Delivery System (Injury, poisoning and procedural complications) | 1 (1) | 0
Elective Surgery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Emesis/Vomiting (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 22 (27) | 0 (0)
Fever (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Lacerations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nausea (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Non-Cardiac Chest Pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Other (Injury, poisoning and procedural complications) | 43 (57) | 0
Pain (Injury, poisoning and procedural complications) | 4 (5) | 0 (0)
Poison Ivy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Swelling (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weakness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Weight Loss (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Arthritis Associated with Spondylitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Digit Injury, Finger/Toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
General - Musculoskeletal Symptoms (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator Cuff Tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Altered Sensorium (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0
Carotid Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive Impairment (Nervous system disorders) | 3 (3) | 0 (0)
Delirium (Nervous system disorders) | 2 (2) | 0 (0)
Dementia (Nervous system disorders) | 5 (5) | 1 (1)
Depression (Nervous system disorders) | 1 (1) | 0 (0)
Dysautonomia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
General - Neurological Symptoms (Nervous system disorders) | 16 (16) | 2 (3)
Hallucinations (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
Speech Difficulty (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 5 (5) | 2 (2)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 3 (3) | 4 (4)
Vaso Vagal Response (Nervous system disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Chronic Obstructive Airway Disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Difficulty Catching Breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Idiopathic Interstitial Lung Diseases (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Disorders (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary Nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
X-ray Finding (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
VASC Hematoma (Vascular disorders) | 2 (2) | 0 (0)
VASC Pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)
Skin Bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal Failure (General disorders) | 0 (0) | 3 (3)
Bacteremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Closed Head Injury (Nervous system disorders) | 0 (0) | 1 (1)
VASC Vessel Dissection (Vascular disorders) | 0 (0) | 1 (1)
Cancer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device/Delivery System (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Elective Surgery (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Fatigue/Generalized Fatigue (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lacerations (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pain Due to a Catheter Drainage Tube (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vessel Stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight Gain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other (Injury, poisoning and procedural complications) | 0 (0) | 13 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are bound by the Abbott Investigator Agreement, which includes confidentiality clauses and limits what study details and data they are permitted to share and/or publish without prior authorization from Abbott.

DOCUMENTS (2):
  • Study Protocol (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT04011722/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT04011722/SAP_001.pdf